CLINICAL TRIAL: NCT04995445
Title: Retrospective Evaluation of the Effect of Ultrasound-guided Obturator Nerve Block on Complications in Transurethral (TUR-M) Resection Surgery for Bladder Side Wall Tumors.
Status: Completed | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, HULYA TOPCU, assistant professor, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2019-158
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Efficacy of Peripheral Nerve Blocks on Complications, Morbidity and Mortality
Keywords: Obturator nerve block; complications of transurethral resection; TUR-M

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the effectiveness of obturator nerve block added to spinal anesthesia in the operation of transurethral resection (TUR-M) of bladder lateral-infrolateral wall tumors on the obturator reflex and related complications was investigated.

ELIGIBILITY:
retrospective study

Inclusion criteria:

* Patients over the age of 18 who have undergone bladder tumor surgery and whose anesthesia method is spinal anesthesia

Exclusion Criteria:

* under 18 years old , received general anesthesia pregnant and pediatric patient data not used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: more than 18 years regional anesthesia method was applied The files of patients who underwent Tur-M surgery were reviewed retrospectively.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Effect of ultrasound-guided obturator nerve block on complications in transurethral resection of bladder cancer | 2 year
  patient who underwent spinal anesthesia and obturator block

SECONDARY OUTCOMES:
Effect of ultrasound-guided obturator nerve block on complications in transurethral resection of bladder cancer | 2 year
  The patient group who underwent spinal anesthesia and obturator block and the group without obturator block

CONTACTS AND LOCATIONS:
Locations (1):
- Çorum training and research state hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided